CLINICAL TRIAL: NCT02532270
Title: Detecting Hypotension By Continuous Non-invasive Arterial Pressure Monitoring During Spinal Anaesthesia for Cesarean Section:A Prospective,Randomized, Controlled Study
Brief Title: Detecting Hypotension By Continuous Non-invasive Arterial Pressure Monitoring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chao Han, Department of Anesthesiology, Department of Obstetrics and Gynecology Hospital, Fudan University, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CNAP 01
Record Dates: First submitted 2015-08-13; First posted 2015-08-25 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Hypotension
Keywords: obstetric; anesthesia; hypotension; arterial pressure; measurement techniques
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group C (Experimental): Arterial pressure of the patients in Group C is measured by continuous non-invasive arterial pressure (CNAP).When systolic blood pressure decreased by over 20% of the basic value or systolic blood pressure lower than 100mmHg after spinal anaesthesia,phenylephrine was administered 50ug .If systolic blood pressure did not improve after 1 minute,phenylephrine was administered repeatedly until systolic blood pressure return to normal.
  Interventions: Drug: phenylephrine
- Group N (Experimental): Arterial pressure of the patients in Group N is measured by intermittent oscillometric non-invasive arterial pressure (NIAP).When systolic blood pressure decreased by over 20% of the basic value or systolic blood pressure lower than 100mmHg after spinal anaesthesia,phenylephrine was administered 50ug .If systolic blood pressure did not improve after 1 minute,phenylephrine was administered repeatedly until systolic blood pressure return to normal.
  Interventions: Drug: phenylephrine

INTERVENTIONS:
Drug: phenylephrine — When systolic blood pressure decreased by over 20% of the basic value or systolic blood pressure lower than 100mmHg after spinal anaesthesia,phenylephrine was administered 50ug in Group C and Group N.If systolic blood pressure did not improve after 1 minute,phenylephrine was administered repeatedly until systolic blood pressure return to normal.
  Other Names: Phenylephrine Hydrochloride

SUMMARY:
The purpose of this study is to determine whether continuous non-invasive arterial pressure (CNAP) monitoring is beneficial to maintain maternal hemodynamic stability and improve the outcomes of maternal and fetal comparing with intermittent oscillometric non-invasive arterial pressure (NIAP)measurement during spinal anaesthesia for cesarean section .

DETAILED DESCRIPTION:
Peri-operative hypotension and fluctuation of arterial blood pressure (BP) during spinal anaesthesia are common. Hypotension causes maternal side-effects such as unconsciousness, dizziness, nausea, and vomiting. The potential fetal side-effects are caused by a reduction in the uterine blood flow with consequent reduced oxygen supply and acidosis reflected by impaired blood gas analyses and impaired Apgar scores. Because of the potential harm to the fetus and the dependency of fetal oxygenation on maternal arterial pressure (AP), it has been strongly recommended to closely monitor mother's arterial pressure and to treat hypotension immediately. Non-invasive arterial pressure (NIAP) measurement is a common method for monitoring in clinical. These hypotension episodes probably would be detected with delay by NIAP measurement on account of its discontinuous. A monitor for continuous non-invasive arterial pressure monitoring (CNAPTM Monitor 500, CNSystems Medizintechnik AG,Graz, Austria) using the volume-clamped method. It can monitor timely and provide beat-to-beat value of arterial pressure.

The purpose of this study is to determine whether continuous non-invasive arterial pressure (CNAP) monitoring is beneficial to maintain maternal hemodynamic stability and improve the outcomes of maternal and fetal.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective caesarean section with spinal anaesthesia
* pregnancy week above 36

Exclusion Criteria:

* age<18 yr
* cardiac arrhythmia
* vascular pathologies of the upper limbs (recent vascular surgery, Raynaud's disease， vascular stenosis)
* contraindication for spinal anaesthesia
* emergency case

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
the maximum change of systolic blood pressure(SBP),assessed using continuous non-invasive arterial pressure device or intermittent oscillometric arterial pressure measurement | between the spinal anesthetic injection and the delivery of the fetus and placenta,assessed up to 30 mins
  (baseline SBP-minimum SBP)/baseline SBP

SECONDARY OUTCOMES:
Detecting the occurrence of hypotension | between the spinal anesthetic injection and the delivery of the fetus and placenta,assessed up to 30 mins
  systolic blood pressure decreased by over 20% of the baseline or systolic blood pressure lower than 100mmHg
Neonatal outcome was assessed with Apgar scores | between the spinal anesthetic injection and the delivery of the fetus and placenta,assessed up to 30 mins
umbilical cord blood gases analysis at birth | between the spinal anesthetic injection and the delivery of the fetus and placenta,assessed up to 30 mins
the incidence of nausea and vomiting on account of hypotension | between the spinal anesthetic injection and the delivery of the fetus and placenta,assessed up to 30 mins
  The presence of nausea and vomiting was measured on a 3-point scale of 1,2, and 3 indicating no nausea and no vomiting, nausea only, and both nausea and vomiting, respectively. Assessments were done at 1-minute intervals after the spinal injection until 25 min.
the incidence of dizziness on account of hypotension | between the spinal anesthetic injection and the delivery of the fetus and placenta,assessed up to 30 mins
  assessment:yes=patient had dizziness,no=patient had no dizziness
the incidence of dyspnea on account of hypotension | between the spinal anesthetic injection and the delivery of the fetus and placenta,assessed up to 30 mins
  assessment:yes=patient had dyspnea,no=patient had no dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Shaoqiang Huang, Dr, Study Director — Department of Anesthesiology, Department of Obstetrics and Gynecology Hospital, Fudan University
Locations (1):
- Department of Anesthesiology, Department of Obstetrics and Gynecology Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Result] Ilies C, Kiskalt H, Siedenhans D, Meybohm P, Steinfath M, Bein B, Hanss R. Detection of hypotension during Caesarean section with continuous non-invasive arterial pressure device or intermittent oscillometric arterial pressure measurement. Br J Anaesth. 2012 Sep;109(3):413-9. doi: 10.1093/bja/aes224. Epub 2012 Jul 12. PMID 22798273
- [Result] Jeleazcov C, Krajinovic L, Munster T, Birkholz T, Fried R, Schuttler J, Fechner J. Precision and accuracy of a new device (CNAPTM) for continuous non-invasive arterial pressure monitoring: assessment during general anaesthesia. Br J Anaesth. 2010 Sep;105(3):264-72. doi: 10.1093/bja/aeq143. Epub 2010 Jul 13. PMID 20627878
- [Result] Banerjee A, Stocche RM, Angle P, Halpern SH. Preload or coload for spinal anesthesia for elective Cesarean delivery: a meta-analysis. Can J Anaesth. 2010 Jan;57(1):24-31. doi: 10.1007/s12630-009-9206-7. Epub 2009 Oct 27. PMID 19859776
- [Result] Lee A, Ngan Kee WD, Gin T. A quantitative, systematic review of randomized controlled trials of ephedrine versus phenylephrine for the management of hypotension during spinal anesthesia for cesarean delivery. Anesth Analg. 2002 Apr;94(4):920-6, table of contents. doi: 10.1097/00000539-200204000-00028. PMID 11916798
- [Result] Maayan-Metzger A, Schushan-Eisen I, Todris L, Etchin A, Kuint J. Maternal hypotension during elective cesarean section and short-term neonatal outcome. Am J Obstet Gynecol. 2010 Jan;202(1):56.e1-5. doi: 10.1016/j.ajog.2009.07.012. Epub 2009 Aug 28. PMID 19716536